CLINICAL TRIAL: NCT01300715
Title: An Alternative Technique for Lumbar Medial Branch Radiofrequency: Comparison With the Empirical Technique
Acronym: MBRF LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Jeeyoun Moon, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBRF
Record Dates: First submitted 2011-01-31; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-10

CONDITIONS: Low Back Pain; Lumbar Facet Joint Pain; Arthropathy
Keywords: zygapophysial joint; facet joint; low back pain; radiofrequency; neurotomy
MeSH Terms: conditions — Low Back Pain; Joint Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MBRF (Active Comparator)
  Interventions: Procedure: lumbar medial branch radiofrequency neurotomy

INTERVENTIONS:
Procedure: lumbar medial branch radiofrequency neurotomy — the classic tunnel vision technique versus the alternative technique

SUMMARY:
In spite that variable techniques for lumbar MBRF exists, the tunnel vision technique is widely recommended for exact radiofrequency needle placement. However, this method uses the concept of a steep caudocephalad axial tilt of the fluoroscopy beam, which result in unusual appearance of vertebral structures and a long distance from skin to the target site. In our institution, therefore, the investigators have used a modified method that is easy and safe to place RF needle parallel to the lumbar medial branch in oblique fluoroscopic view.

Accordingly, our objectives were to evaluate our modified technique for lumbar MBRF, comparing with the tunnel vision technique, and additionally to assess complications with respect to these two techniques.

DETAILED DESCRIPTION:
The zygapophysial (facet) joint pain has been a challenging condition for pain specialists since the 20th century. According to the previous reports, degenerative changes of facet joint account for 10% - 15% of the cases with chronic low back pain. However, it is a major source of frustration that there is no definitive standard to document a clinical diagnosis and few validated treatment about lumbar facet joint pain.

Although it has been a subject of debate how best to select patients, radiofrequency (RF) neurotomy is frequently performed procedure for patients with lumbar facet generated pain. Lumbar medial branch radiofrequency (MBRF) is assumed to be effective and safe treatment for lumbar facet joint pain with 1.0% rate of minor complications per lesion site. The rationale and efficacy of lumbar MBRF would depend on the use of meticulous radiofrequency (RF) needle placement with stringent patient selection.

In spite that variable techniques for lumbar MBRF exists, the tunnel vision technique is widely recommended for exact RF needle placement. However, this method uses the concept of a steep caudocephalad axial tilt of the fluoroscopy beam, which result in unusual appearance of vertebral structures and a long distance from skin to the target site. In our institution, therefore, the investigators have used a modified method that is easy and safe to place RF needle parallel to the lumbar medial branch in oblique fluoroscopic view.

Accordingly, our objectives were to evaluate our modified technique for lumbar MBRF, comparing with the tunnel vision technique, and additionally to assess complications with respect to these two techniques.

ELIGIBILITY:
Inclusion Criteria:

- Chronic low back pain patients (pain duration > 6 months) who had not responded to previous treatment, underwent screening medial branch blocks (MBBs) using 0.5% levobupivacaine hydrochloride (Chirocaine®, Abbott Korea Ltd, Seoul, Republic of Korea) 0.5 mL at each of the standard target points.8 Patients that achieved at least 80% pain relief by screening MBBs underwent controlled comparative local anesthetic blocks using 1% lidocaine (0.5 mL) and 0.5% levobupivacaine (0.5 mL). Those that achieved greater than 80% pain relief following double blocks were eligible for lumbar MBRF, but those with prolonged responses to screening or dual-controlled comparative MBBs were not considered eligible.

Exclusion Criteria:

1. Duration of low back pain < 6 mo
2. Single diagnostic block
3. Prolonged responses to screening or dual-controlled comparative MBBs
4. Discogenic pain verified by controlled discography
5. Evidence of radiculopathy, as determined by history, physical examination, and radiologic studies
6. Structural lumbar spinal deformity
7. Rapidly worsening pain, numbness, weakness, hyperreflexia, changes in bladder function, and other neurological symptoms which should prompt a reevaluation and surgical evaluation.
8. Previous back surgery
9. Severe psychiatric illness

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale (NRS)(1) | change from baseline in NRS at 4 weeks
  Preprocedure low-back pain recorded on a 0 to 10 numerical rating scale (NRS)versus NRS at one-month follow-up visits

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI)(1) | change from baseline in ODI at 4 weeks
  Preprocedure Oswestry Disability Index (ODI) versus ODI at one-month follow-up visit
time to complete the procedures | on procedure
  Time required to complete each procedure (skin-to-lesion time, separately)
7-point global perceived effect (GPE) scale about low back pain (1) | change from baseline in GPE scale at 4 weeks after the procedure
  1. = worse than ever
  2. = much worsened
  3. = slightly worsened
  4. = unchanged
  5. = slightly improved
  6. = much improved
  7. = completely recovered
Complication (1) | at one-month follow-up visit
  Complications associated to the procedures
  1. localized pain at radiofrequency sites
  2. neuritic pain
  3. a new sensory or motor deficit
  4. others
medication reduction (1) | baseline and 4 weeks
  doses of preprocedural analgesics versus postprocedural medication reduction
NRS(3) | Change from baseline in NRS at 12 weeks
  preprocedural low back pain recorded on a 0 to 10 numerical rating scale versus NRS at a 3-month follow-up visit
procedure-related pain of numerical rating scale (NRS) | after 10 minutes following the procedure
  Procedure-related pain as determined by NRS is recorded immediately after lumbar medial branch radiofrequency.
Oswestry Disability Index (ODI)(3) | change from baseline in ODI at 12 weeks
  Preprocedure Oswestry Disability Index (ODI) versus ODI at three-month follow-up visit
7-point global perceived effect (GPE) scale about low back pain (3) | change from baseline in GPE scale at 12 weeks after the procedure
  1. = worse than ever
  2. = much worsened
  3. = slightly worsened
  4. = unchanged
  5. = slightly improved
  6. = much improved
  7. = completely recovered
Complication (3) | at three-month follow-up visit
  Complications associated to the procedures
  1. localized pain at radiofrequency sites
  2. neuritic pain
  3. a new sensory or motor deficit
  4. others
medication reduction (3) | baseline and 12 weeks
  doses of preprocedural analgesics versus postprocedural medication reduction
Volume of local anesthetic | on procedure
  Volume of local anesthetic required for superficial and deep anesthesia, separately

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Sungnam, Kyonggi-do, South Korea